CLINICAL TRIAL: NCT06782568
Title: Avoidance of Insulin-induced Lipohypertophy in People With Diabetes: A Feasibility Study of Implementation of Ultrasound Scanning Within Diabetes Clinics
Brief Title: Avoidance of Insulin-induced Lipohypertophy in People With Diabetes Using Ultrasound Scanning Within Diabetes Clinics
Acronym: Avoid-Lipo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Edge 175976; WREE_PA7435 (Other Grant/Funding Number: The NIHR Imperial Biomedical Research Centre (BRC))
Record Dates: First submitted 2025-01-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes (T1D); Type 2 Diabetes, Insulin Requiring
Keywords: Lipohypertophy; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Single arm non-randomised feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound scanning of insulin injection sites (Experimental): Participants will undergo clinical examination followed by ultrasound scanning (USS) of the injection sites at baseline. If there is no significant lipohypertophy (LH) detected by USS, participants will take no further part in the study. If there is LH detected on USS, an individualised map of LH sites and clear sites will be drawn, and the participant will be asked to avoid LH sites for the next 6 months. Follow up remote/virtual/F2F visits will be conducted at 1 and 3 months. The final visit at 6 months will consist of a repeat clinical examination followed by a repeat USS.
  Interventions: Diagnostic Test: Ultrasound Scan

INTERVENTIONS:
Diagnostic Test: Ultrasound Scan — Participants will undergo an ultrasound scan of insulin injection sites at baseline and after 6 months.

SUMMARY:
Diabetes is a common long-term health condition globally. Type 1 diabetes requires insulin treatment right from diagnosis. Similarly, many living with type 2 diabetes eventually require insulin injections as the condition progresses. A common but often underappreciated complication associated with insulin use is the formation of fatty tissue at injection sites, known as "Lipos," a shorthand for "Lipohypertrophy." These Lipos can interfere with insulin absorption, leading to an altered insulin action profile. This results in glucose fluctuations increasing the risk of both high and low glucose levels.

In current medical practice, Lipos are assessed through clinical examination, specifically by physically palpating the injection sites. Research indicates that approximately 40% of insulin-treated individuals may have Lipos. However, manual palpation can often overlook these fatty deposits. Ultrasound scanning (USS) presents a more effective method for detecting Lipos. Studies that have employed ultrasound scanning have reported a much higher prevalence, reaching up to 86%.

The primary goal of this study is to ascertain whether the avoidance of ultrasound-identified Lipos can improve glucose regulation. The focus will be on individuals using continuous glucose monitoring who exhibit high glucose fluctuations and less time within their target range. By focusing on this population, the chances of identifying those with Lipos will increase.

Participants will undergo a clinical examination followed by an ultrasound scan. Those found to have Lipos will receive guidance on avoiding those sites and education on insulin injection techniques. Glucose data will be collected periodically over the next 24 weeks. After this period, participants will return for a follow-up ultrasound scan. Additionally, members of the diabetes care team will be trained to conduct the ultrasound scans. Data from this study may also be utilized to develop artificial intelligence algorithms aimed at identifying Lipos in future ultrasound scans.

DETAILED DESCRIPTION:
This will be a single-centre, prospective, open-label, non-randomized feasibility study. Participants will be recruited through diabetes clinics at Imperial College Healthcare NHS Trust, London, UK. Written informed consent will be obtained.

Key Inclusion criteria:

* Any diabetes treated with either multiple daily injection therapy (MDI) or an insulin pump (including automated insulin delivery systems), currently using any form of continuous glucose monitoring (CGM) with use >70% in the last 4 weeks. (Those with type 2 diabetes MDI is defines as more than one insulin injection per day)
* No anticipated changed to diabetes treatment in the next 6 months.
* The coefficient of variation (CV) of CGM glucose >36% and Time in the range between 3.9 to 10.0 mmol/l is <70%
* Willing to undergo a clinical examination and USS for detection of LH sites

Exclusion criteria:

* Any other physical disease or people with known severe mental illness that are likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Estimated Glomerular Filtration Rate (e-GFR) < 25
* Known to have any form of lipodystrophy disorder either primary or secondary to other medical conditions
* Dercum's disease
* Women who are pregnant or planning pregnancy
* The participant has an active major life-threatening illness limiting the participants life-expectancy to <6 months

The study will be conducted at Imperial College Healthcare NHS Trust. All consented participants will enter a 2-week run-in period where baseline demographic data will be collected and baseline clinical examination and USS will be performed. Continuous glucose monitoring (CGM) data from patients own CGM device will be collected and HbA1c test performed if not done within last 2 weeks. A map of Lipo site will be created and participant advised to avoid these sites for next 24 weeks. CGM data at 4 weeks and 12 weeks post-baseline USS scan will be collected either remotely or in-person. End of study USS, CGM data collection and HbA1c will be conducted at 24 weeks after the baseline USS.

Details of study visits:

Visit 1: Screening & Enrolment

Potentially eligible participants will attend the diabetes clinic or clinical research facility or will be seen during their scheduled clinic appointments as preferred by participants and availability of clinical space. Following written informed consent, baseline clinical data will be collected from all participants. Information sheets will be provided in advance to potential participants. Following informed consent, those interested in participating will be assessed to determine if they meet the inclusion criteria listed above. A blood sample will be taken for HbA1c & kidney function if no result is available within the last two weeks. Women of childbearing potential will have a βHCG test to exclude pregnancy.

The following data will be recorded in the CRF:

1. Informed consent obtained
2. General Clinical

   1. Date of Birth
   2. Gender
   3. Weight and height
   4. Non-diabetes related co-morbidities
3. Diabetes clinical

   1. Date of diagnosis
   2. Duration of insulin therapy
   3. Insulin dose (including average total daily insulin, average daily basal insulin, average daily bolus insulin) and other diabetes medications
   4. Complication status
   5. History of severe hypoglycaemia - coma or convulsion (events requiring assistance for recovery in the past 12 months)
   6. History of diabetic ketoacidosis or non-ketotic hyperosmolar coma in the last 12 months
   7. History of participation in structured education or virtual education
   8. Number of boluses per day & Any evidence of missed boluses
   9. Carbohydrate counting method and use of dynamic insulin doses for meals and corrections
   10. In females, menstrual history and history of high glucose and or glucose variability around periods

CGM data Glucose data from the CGM device will be downloaded and stored in an approved computer. Summary CGM statistics using usual clinical software (Carelink, Libreview, Dexcom Clarity) will also be recorded for last 4 weeks.

Visit 2: Baseline Ultrasound Scan (USS)

Participants will have a clinical examination of the insulin injection sites followed by USS of the injection sites. Findings will be documented in the case report forms, and individual maps of injection sites with Lipos created, and participants will be advised to avoid Lipo sites for the next 24 weeks. Insulin needle lengths (4 mm needles advised if on longer needles) and injection techniques will also be paid attention to.

If no significant lipohypertophy (LH) is detected by USS, participants will take no further part in the study

Visit 3: Four-week follow visit

This visit could be done as a remote visit. Glucose data from the CGM device will be downloaded and stored. Summary CGM statistics using usual clinical software (Carelink, Libreview, Dexcom Clarity) will also be recorded for last 4 weeks.

Visit 4: 12-week follow visit

This visit could be done as a remote visit. Glucose data from the CGM device will be downloaded and stored. Summary CGM statistics using usual clinical software (Carelink, Libreview, Dexcom Clarity) will also be recorded for last 4 weeks.

Visit 5: End of Study Visit (24-weeks)

All participants will have blood sample taken for HbA1c. Glucose data from the CGM device will be downloaded and stored. Summary CGM statistics using usual clinical software (Carelink, Libreview, Dexcom Clarity) will also be recorded for last 4 weeks. Participants will have a clinical examination of the insulin injection sites followed by USS of the injection sites. Information about current insulin doses will also be collected. This will be the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Any type of diabetes of at least 1-year duration managed with multiple daily injections (MDI [ie separate rapid-acting and basal insulin injections]) or insulin pump therapy (CSII)
* Currently using any form of continuous glucose monitoring (CGM) with use >70% in the last 4 weeks
* No anticipated changes to diabetes treatment in the next 6 months such as introduction of novel agents like GLP-1, SGLT2 or introduction (Tupe 2 diabetes) or AID (Type 1 diabetes)
* Coefficient of variation (CV) of CGM glucose >36% and Time in the range between 3.9 to 10.0 mmol/l is <70%
* The participant is willing and able to implement the study requirements and undergo two ultrasound scans of the insulin injection sites
* Participants is able understand English sufficiently for safe study conduct

Exclusion Criteria:

* Any other physical disease or people with known severe mental illness that are likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Known to have any form of lipodystrophy disorder either primary or secondary to other medical conditions
* Dercum's disease
* Women who are pregnant or planning pregnancy
* The participant has an active major life-threatening illness limiting the participants life-expectancy to <6 months
* Estimated Glomerular Filtration Rate (e-GFR) < 25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Time in Range (3.9 to 10.0 mmol/l) | From enrollment to the end of treatment at 24 weeks
  Time spent in the target glucose range between 3.9 to 10.0 mmol/l (70 to 180 mg/dl) based on sensor glucose levels for the last 4 weeks of the 24 week study period

SECONDARY OUTCOMES:
HbA1c | From enrollment to the end of treatment at 24 weeks
  Change in HbA1c from baseline
Mean glucose | From enrollment to the end of treatment at 24 weeks
  Mean glucose levels at 24 weeks
Time above range (Level 1) | From enrollment to the end of treatment at 24 weeks
  Time spent above target glucose (10.0 mmol/l) (180 mg/dl) (Level 1 hyperglycaemia)
Time above range (Level 2) | From enrollment to the end of treatment at 24 weeks
  Time spent above target glucose (13.9 mmol/l) (250 mg/dl) (Level 2 hyperglycaemia)
Time below range (Level 1) | From enrollment to the end of treatment at 24 weeks
  Time spent below target glucose (<3.9mmol/l) (<70mg/dl) (Level 1 hypoglycaemia)
Time below range (Level 2) | From enrollment to the end of treatment at 24 weeks
  Time spent below target glucose (<3.0mmol/l) (<54mg/dl) (Level 2 hypoglycaemia)
Insulin doses | From enrollment to the end of treatment at 24 weeks
  Average total daily insulin dose, basal and bolus dose
Severe Hypoglycaemia | From enrollment to the end of treatment at 24 weeks
  Frequency of severe hypoglycaemic episodes as defined by the American Diabetes Association
Resolution of Lipohypertrophy (LH) | From enrollment to the end of treatment at 24 weeks
  Resolution rate of Lipohypertrophy (% of participants affected and number of distinct LH sites per participant)
Time in Range (3.9 to 10.0 mmol/l) | From enrollment to the end of treatment at 12 weeks
  Time spent in the target glucose range between 3.9 to 10.0 mmol/l (70 to 180 mg/dl) based on sensor glucose levels
Time in Range (3.9 to 10.0 mmol/l) | From enrollment to the end of treatment at 4 weeks
  Time spent in the target glucose range between 3.9 to 10.0 mmol/l (70 to 180 mg/dl) based on sensor glucose levels
Glucose variability | From enrollment to the end of treatment at 24 weeks
  Coefficient of Variation of glucose levels at 24 weeks

OTHER OUTCOMES:
Adverse Events | From enrollment to the end of treatment at 24 weeks
  Adverse events will be tabulated and reported

CONTACTS AND LOCATIONS:
Overall Officials: Lalantha Leelarathna, PhD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a single-arm feasibility study.

REFERENCES:
- [Background] Mader JK, Fornengo R, Hassoun A, Heinemann L, Kulzer B, Monica M, Nguyen T, Sieber J, Renard E, Reznik Y, Rys P, Stozek-Tutro A, Wilmot EG. Relationship Between Lipohypertrophy, Glycemic Control, and Insulin Dosing: A Systematic Meta-Analysis. Diabetes Technol Ther. 2024 May;26(5):351-362. doi: 10.1089/dia.2023.0491. Epub 2024 Feb 12. PMID 38215209